CLINICAL TRIAL: NCT01300065
Title: A Study to Evaluate the Product Performance of Two Daily Disposable Contact Lenses
Brief Title: Evaluation of Two Daily Disposable Contact Lenses.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 642
Record Dates: First submitted 2011-02-17; First posted 2011-02-21 (Estimated); Results first posted 2020-10-06 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-09

CONDITIONS: Myopia
Keywords: contact lens
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental- Soflens (Experimental): Bausch & Lomb experimental soflens daily disposable contact lens packaged in an investigational storage solution.
  Interventions: Device: Experimental- Soflens
- Marketed - Soflens (Active Comparator): Bausch & Lomb daily disposable marketed soflens contact lens packaged with: 0.5% poloxamine in buffered saline solution.
  Interventions: Device: Marketed - Soflens

INTERVENTIONS:
Device: Experimental- Soflens — A new pair of lenses will be worn each day while the subject is in the study
  Arms: Experimental- Soflens
Device: Marketed - Soflens — A new pair of lenses will be worn each day while the subject is in the study.
  Arms: Marketed - Soflens

SUMMARY:
The objective of this clinical study is to evaluate the product performance of SofLens daily disposable contact lenses packaged in the investigational Test solution versus SofLens daily disposable contact lenses packaged in Control, solution as it relates to comfort when used by subjects who use technology devices (eg, Personal Digital Assistants [PDAs], computers, electronic game consoles, hand-held electronic devices, electronic book readers, etc) on an average of 4 hours per day over a week's time for a minimum of 4 days each week.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be correctable through spherocylindrical refraction to 32 letters (0.3 logMAR) or better (distance, high contrast) in each eye.
* Subjects must be free of any anterior segment disorders.
* Subjects must be adapted soft contact lens wearers and wear a lens in each eye and each lens must be of the same manufacture and brand.
* Subjects must be myopic and require contact lens correction from -0.50 D to -6.00 D in each eye.
* Subjects must be willing and able to wear the study lenses for at least 8 hours (12 hours or more is recommended) each day throughout the duration of the study.
* Subjects must use a technologic device for an average of 4 hours per day over a week's time and at a minimum of 4 days per week.

Exclusion Criteria:

* Subjects who have worn gas permeable (GP) contact lenses within the last 30 days or who have worn polymethylmethacrylate (PMMA) lenses within the last three months.
* Subjects with any systemic disease currently affecting ocular health or which in the Investigator's opinion may have an effect on ocular health during the course of the study.
* Subjects using any systemic or topical medications that will, in the Investigator's opinion, affect ocular physiology or lens performance.
* Subjects with an active ocular disease or who are using any ocular medication.
* Subjects with corneal infiltrates, of ANY GRADE, are not eligible.
* Subjects with any "Present" finding during the slit lamp examination that, in the Investigator's judgment, interferes with contact lens wear.
* Subjects with any scar or neovascularization within the central 4 mm of the cornea.
* Subjects who have had any corneal surgery (eg, refractive surgery).
* Subjects who are allergic to any component in the study care products.
* Subjects may not use their habitual rewetting drops while participating in this study.

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 441 (Actual)
Dates: Start 2011-01; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beverly J Barna, CCRA, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb Incorporated, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 441 participants (882 eyes) enrolled, 221 in the test group and 220 in the control group. There were 434 eligible participants (868 eyes) who participated in the study, 216 in the test group and 218 in the control group.
Period: Overall Study
Arm/Group | Experimental- Soflens | Marketed - Soflens
Started | 221 | 220
Completed | 215 | 217
Not Completed | 6 | 3

BASELINE CHARACTERISTICS:
Population: Eligible, dispensed participants were summarized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental- Soflens | Marketed - Soflens | Total
Number analyzed (Participants) | 215 | 216 | 431
Age, Continuous [Mean (Full Range); unit: years] | 27.1 [15 to 40] | 26.6 [15 to 50] | 26.8 [15 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 153 | 293
  Male | 75 | 63 | 138

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eyes With > Grade 2 Slit Lamp Findings
Description: Graded slit lamp findings for each eye, including epithelial edema, epithelial microcysts, corneal staining, limbal and bulbar injections, upper lid tarsal conjunctival abnormalities, corneal neovascularization, and corneal infiltrates were graded for severity on a scale from 0 (No Finding) to 4 (Severe Finding). The outcome measure is any finding > grade 2, across abnormalities.
Time Frame: 2 weeks
Population: There were 438 eyes in the test group and 434 eyes in the control group that were assessed for this outcome measure.
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Experimental- Soflens | Marketed - Soflens
Number analyzed (Participants) | 219 | 217
Number analyzed (eyes) | 438 | 434
eyes | 0 | 0

2. Secondary Outcome: Initial Lens Performance Survey
Description: A lens performance survey was given to each participant at the Screening/Dispensing Visit, three minutes following insertion of the study lenses. Lens performance was assessed by eye for the following parameters: burning/stinging upon insertion, comfort upon insertion, ease of handling/insertion, vision upon insertion, and lens cleanness upon insertion. As with symptoms/complaints, responses were on a scale from 0 to 100, with 0 being the most unfavorable score.
Time Frame: At dispensing
Population: There were 426 eyes in the test group and 424 eyes in the control group that were assessed for this outcome measure.
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Experimental- Soflens | Marketed - Soflens
Number analyzed (Participants) | 213 | 212
Number analyzed (eyes) | 426 | 424
score on a scale
  Burning/stinging upon insertion | 91.6 (18.7) | 91.0 (18.7)
  Comfort Upon Insertion | 83.8 (21.1) | 83.9 (21.2)
  Ease of Handling/Insertion | 77.2 (26.2) | 79.4 (26.3)
  Vision Upon Insertion | 89.3 (15.5) | 88.4 (15.6)
  Lens Cleanness Upon Insertion | 95.4 (10.8) | 94.9 (10.9)

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Adverse events were not coded. Therefore, source vocabulary is not applicable.There were 440 eyes dispensed test lenses and 436 eyes dispensed control lenses, assessed for adverse events.
Arm/Group | Experimental- Soflens | Marketed - Soflens
Serious Adverse Events (participants affected / at risk) | 0/221 | 0/220
Other Adverse Events (participants affected / at risk) | 0/221 | 0/220

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.